CLINICAL TRIAL: NCT05979727
Title: Double-blind, Randomized, Dose-response Study of RE02 in Healthy Subjects
Brief Title: Dose-finding PKPD Trial for RE02 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was closed due to futility
Sponsor: Reconnect Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: MEO-DMT-VR
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Manitol
- Low dose of RE02 (Active Comparator)
  Interventions: Drug: RE02
- Moderate dose of RE02 (Active Comparator)
  Interventions: Drug: RE02
- High dose of RE02 (Active Comparator)
  Interventions: Drug: RE02

INTERVENTIONS:
Drug: RE02 — Low, medium or high dose of RE02
  Arms: High dose of RE02; Low dose of RE02; Moderate dose of RE02
Drug: Manitol — Placebo Comparator
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare corresponding inter- and intraindividual pharmacokinetic and pharmacodynamic profiles including assessments of safety & tolerability of three different doses against a placebo control.

DETAILED DESCRIPTION:
Participants will undergo a series of four study days with varying doses of RE02 and a placebo. The intervention is embedded in controlled environment and continuous psychological support. Pharmacokinetic and pharmacodynamic assessments are obtained over the course of 6 hours on each study visit to estimate dose-exposure relationship and drug-drug-interaction. Additionally, the occurrence of adverse events will be closely monitored throughout the whole study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable to give informed consent for the participation in the study after it has been thoroughly explained
* Willing to refrain from drinking alcohol one day before testing days and caffeinated drinks at the testing days and from consuming psychoactive substances or other medications for 2 weeks before testing days and for the duration of the study
* Already experienced with psychedelic substances (at least 5 prior experiences - microdoses do not count)
* Able and willing to comply with all study requirements
* Informed consent form was signed
* Good knowledge of the German language
* Participant informs study physicians / project scientists about simultaneous treatment or therapy with other physicians and about current intake of psychotropic substances or medication
* Women of childbearing potential are required to use effective, established contraception, such as oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Exclusion Criteria:

* Previous significant adverse response to a hallucinogenic drug
* Participation in another study where pharmaceutical compounds will be given
* Presence of Axis I affective, anxiety, or dissociative disorders
* Present or antecedent diagnosis of bipolar disorder (I, II, not otherwise specified), schizophrenia, schizoaffective disorder, psychosis, or other disorders from the psychotic spectrum
* First-degree relatives with present or antecedent schizophrenia, schizoaffective disorder, or bipolar disorder type I
* History of head trauma, seizures, cancer, or cerebrovascular accidents
* Recent cardiac or brain surgery
* Current abuse of medication or psychotropic substances (including nicotine addiction) according to SCID I criteria
* Presence of major internal or neurological disorders (including sepsis, pheochromocytoma, thyrotoxicosis, drug-induced fibrosis, familiar or basilar artery migraine)
* Cardiovascular disease (hypertonia, coronary artery disease, heart insufficiency, myocardical infarction, coronary spastic angina)
* Peripheral vascular disease (thromboangiitis obliterans, luetic arteritis, severe arteriosclerosis, thrombophlebitis, Raynaud's disease)
* Cerebrovascular disease (e.g., stroke, intracranial bleeding / hemorrhage, intracranial aneurysm)
* Serious abnormalities in ECG or blood count/chemistry
* Liver or renal or pulmonary disease
* Current use of medications with significant interaction potential with MAOI (e.g., antidepressants, antipsychotics, psychostimulants, dopaminergic/serotonergic agents, anticonvulsants)
* high risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, serious current stressors, lack of social support)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter "Cmax" | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes in Cmax of several doses of RE02
Pharmacokinetic parameter "Area under the curve (AUC)" | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes in AUC of several doses of RE02.
Pharmacokinetic parameter "T1/2" | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes in T1/2 of several doses of RE02.
Incidence of Treatment-Emergent Adverse Events | On study days 1,2,3,4
  Dose-dependent changes in incidence of adverse drug reactions
Blood count (Lab biochemistry) | Changes from baseline to End of Study, an average of 4 weeks
  Changes from baseline in blood count
Clinical chemistry (Lab biochemistry) | Changes from baseline to End of Study, an average of 4 weeks
  Changes from baseline in any clinical chemistry parameter with potential clinical relevance.
Blood coagulation (Lab biochemistry) | Changes from baseline to End of Study, an average of 4 weeks
  Changes from baseline in blood coagulation
QT interval (12-lead Electrocardiogram [ECG]) | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes of QT intervals assessed by clinical 12-lead ECG)
Blood pressure | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes in systolic and diastolic blood pressure
Heart rate | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes in heart rate
Temperature | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes in temperature
Subjective effects | Changes from baseline to study days 1,2,3,4
  Dose-dependent changes in trajectories of subjective effects

CONTACTS AND LOCATIONS:
Overall Officials: Erich Seifritz, Prof, Principal Investigator — University Hospital of Psychiatry Zurich
Locations (1):
- University Hospital of Psychiatry Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan available to date.